CLINICAL TRIAL: NCT06023914
Title: Analysis of the Effect of Neuromuscular Electro-stimulation on the Performance of Isometric Rotator Cuff Strength in Patients With Tendinopathy.
Brief Title: Analysis of the Effect of Neuromuscular Electro-stimulation on the Performance of Isometric Rotator Cuff Strength.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Pedro Vieira Malachias, Physical Therapist, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ANEEM MRT
Record Dates: First submitted 2023-08-23; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Rotator Cuff Impingement Syndrome; Rotator Cuff Tendinitis; Subacromial Impingement Syndrome
Keywords: shoulder pain; rotator cuff strength
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: The model of strength assessments will be performed randomly. After the individual has performed the first evaluation, he will be evaluated in sequence with the other technique.
Who Masked: Outcomes Assessor
Masking Description: The physiotherapist responsible for carrying out the strength assessments will be blind to which patient has the pathological condition and who is the healthy individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric strength evaluation with a device of electro-stimulation (Experimental): The measurement of rotator cuff strength (medial and lateral rotation) and shoulder elevation will be performed with a Medeor® manual dynamometer. To measure the strength of the medial and lateral rotators, the subject will be positioned in dorsal decubitus, with the shoulder abducted at 45º and in 30º of horizontal adduction (scapular plane), elbow flexed at 90º and neutral rotation, with the dynamometer positioned, respectively, over the distal radio-ulnar joint on the volar or dorsal surface. In all these strength assessments, individuals will be required to perform a maximum isometric contraction for 5 seconds.
  According to the order of randomization, one of the two evaluations will be carried out initially. We will call the evaluation with electrostimulation experimental here. The device to be used will be a GLOBUS® brand equipment, the equipment presents several types of pre-programmed currents, parameters have also been used in similar studies.
  Interventions: Other: STRENGTH EVALUATION WITH ELECTROSTIMULATOR
- Isometric strength evaluation (Active Comparator): The measurement of rotator cuff strength (medial and lateral rotation) and shoulder elevation will be performed with a Medeor® manual dynamometer. To measure the strength of the medial and lateral rotators, the subject will be positioned in dorsal decubitus, with the shoulder abducted at 45º and in 30º of horizontal adduction (scapular plane), elbow flexed at 90º and neutral rotation, with the dynamometer positioned, respectively, over the distal radio-ulnar joint on the volar or dorsal surface. In all these strength assessments, individuals will be required to perform a maximum isometric contraction for 5 seconds.
  We will call this intervention active comparator, as both groups of patients will undergo this evaluation, which will be performed without electrostimulation.
  Interventions: Other: STRENGTH EVALUATION WITHOUT ELECTROSTIMULATOR

INTERVENTIONS:
Other: STRENGTH EVALUATION WITH ELECTROSTIMULATOR — Evaluation of isometric strength using an electrostimulator.
  Arms: Isometric strength evaluation with a device of electro-stimulation
Other: STRENGTH EVALUATION WITHOUT ELECTROSTIMULATOR — Evaluation of isometric strength not using an electrostimulator.
  Arms: Isometric strength evaluation

SUMMARY:
Introduction: Shoulder disorders are a common musculoskeletal problem causing pain and functional loss in different populations. Tendinopathies are a group of pathologies commonly diagnosed in patients with shoulder pain. Weakness of the rotator cuff musculature has already been documented in other studies, evidence in the literature suggests that patients with tendinopathies demonstrate decreased muscle activation, this is caused by pain, changes in nervous system processing and apparently also by structural processes that occur in the tendon .Treatment often involves resistance, isometric exercises aimed at altering pain and restoring function. Some studies have been investigating the use of ENMS (neuromuscular electrical stimulation) in patients undergoing surgical procedures on the shoulder, other studies have also investigated its use in tendinopathies of the lower limbs, as an effective way to decrease inhibition. Objective: The main objective of this study will be to analyze the muscle strength of internal and external rotation of symptomatic shoulders compared to asymptomatic ones when exposed to neuromuscular electrostimulation, associating muscle strength with joint function. Methodology: This will be a cross-sectional study. An expected total of 48 subjects will be divided into two groups, n=24 with tendinopathy of the rotator cuff, confirmed by clinical diagnosis and nuclear magnetic resonance imaging, the other group being healthy individuals, with no history of shoulder pain. These individuals will be evaluated by a first evaluator who will perform the eligibility of the subjects and collect the initial information, the second evaluator will perform the isometric strength evaluation with a manual dynamometer. Two batteries of tests will be performed in both groups, a conventional assessment of isometric strength and the other subject will be submitted to neuromuscular electrostimulation. These strength values in Kgf were normalized for each individual, being divided by the body mass index (BMI) and multiplied by 100, as already performed in previous studies. Expected results: The initial hypothesis is that patients who present with the studied condition when submitted to the strength test with muscular electrostimulation will demonstrate greater isometric strength than when they were tested without the device.

ELIGIBILITY:
Inclusion Criteria:

* Complaint of shoulder pain for at least 30 days
* Age between 25 and 50 years
* Diagnosis of rotator cuff tendinopathy (Jobe, Neer, Hawkins-Kennedy and resisted external rotation test, at least 3 positive tests)
* Magnetic resonance imaging with findings corresponding to rotator cuff tendinopathy?

Inclusion criteria in the health subjects :

* No history of shoulder pain at some point in life
* Age between 25 and 50 years
* Diagnostic Tests for Rotator Cuff Tendinopathy (Jobe, Neer, Hawkins-Kennedy, and resisted external rotation test) NEGATIVE

Exclusion Criteria:

* Contraindications to the use of electrostimulation
* Pregnancy
* History of shoulder, cervical, or thoracic surgery
* Shoulder dislocation
* Fracture
* Labral laceration
* Rheumatic disease
* Complete or partial tear of the rotator cuff
* adhesive capsulitis

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
isometric muscle strength of rotator cuff muscles | short term, immediately after use.
  The primary objective will be to evaluate the isometric muscle strength of the rotator cuff muscles, comparing with the use of the electrostimulator, the measures will be in kgf.

SECONDARY OUTCOMES:
Analyses of isometric strength between groups of healthy and unhealthy individuals. | short term, immediately after use.
  - To analyze isometric external and internal rotator strength relationships between groups of healthy and unhealthy individuals, the measures will be in kgf..
Intra-group group analyses | short term, immediately after use.
  To analyze intra-group isometric external and internal rotator strength relationships, comparing symptomatic and asymptomatic sides, dominant and non-dominant sides, the measures will be in kgf.
other rotator cuff muscle strength analyses | short term, immediately after use.
  To analyze the effect of neuromuscular electrostimulation during the production of isometric strength of external and internal rotators of the shoulder, making comparisons between groups, intra groups, in healthy and unhealthy individuals, the measures will be in kgf.
strength relationship between symptomatic and asymptomatic | short term, immediately after use.
  Analyze the strength relationship between asymptomatic individuals by making comparisons between the symptomatic and asymptomatic sides., the measures will be in kgf.
relationship between symptomatic and asymptomatic and force production | short term, immediately after use.
  To explore the relationships between isometric force production and reproduction of shoulder symptoms or discomfort in symptomatic and asymptomatic individuals., the measures will be in kgf and pain, wich will use the Visual Analog Score for pain.
relationship between symptomatic and asymptomatic and force production and pain | short term, immediately after use.
  To explore the relationships between isometric force production and reproduction of shoulder symptoms or discomfort in symptomatic and asymptomatic individuals., the measures will be in kgf and correlated with pain, wich will use the Visual Analog Score for pain.
relationship between symptomatic and asymptomatic strength and function | short term, immediately after use.
  Observe the relationship between shoulder function and rotator cuff muscle strength in patients with the studied condition, assessed with a scale.
relationship between symptomatic and asymptomatic strength and pain | short term, immediately after use.
  Observe the relationship between shoulder function and rotator cuff muscle strength in patients with the studied condition, assessed with a scale and pain.

IPD SHARING:
Plan to Share IPD: Undecided
I will analyze each request and analyze later